CLINICAL TRIAL: NCT05592613
Title: ID Cap System: Next Generation Ingestible Sensors for Medication Adherence Measurement
Brief Title: Next Generation Ingestible Sensors for Medication Adherence Measurement
Acronym: NextGen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Fenway Institute (Other)
Responsible Party: Principal Investigator, Peter R Chai MD, Emergency Medicine Physician, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022P002497
Record Dates: First submitted 2022-10-12; First posted 2022-10-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: HIV Infection; Adherence, Medication; Adherence, Treatment; Pre-Exposure Prophylaxis; Antiretroviral Therapy
Keywords: Digital Pill System; Pre-Exposure Prophylaxis; Antiretroviral Therapy; Adherence
MeSH Terms: conditions — HIV Infections; Medication Adherence; Treatment Adherence and Compliance | interventions — Drug Delivery Systems; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Pre-Exposure Prophylaxis; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: For 30 days, the next-generation Reader and ID-Cap System will be used in an open-label, observational trial with N=30 participants (N=15 HIV-negative individuals on PrEP and N=15 PLWH on ART).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PrEP Participants (Experimental): Participants will ingest one Truvada digital pill as PrEP per day, for 30 days total, while using the next-generation Reader and ID-Cap System.
  Interventions: Device: Next-generation Reader and ID-Cap System; Drug: Truvada for pre-exposure prophylaxis (PrEP)
- ART Participants (Experimental): Participants will ingest one Biktarvy digital pill as ART per day, for 30 days total, while using the next-generation Reader and ID-Cap System.
  Interventions: Device: Next-generation Reader and ID-Cap System; Drug: Biktarvy for antiretroviral therapy (ART)

INTERVENTIONS:
Device: Next-generation Reader and ID-Cap System — The digital pill system (DPS) is comprised of an ingestible radiofrequency emitter, integrated into a standard gelatin capsule, which then over-encapsulates the study medication (PrEP or ART). On ingestion, the radiofrequency emitter is activated by chloride ions in the stomach, projecting a signal approximately three feet off the body. This radio signal is acquired by a wearable device (Reader) which stores and forwards data to a smartphone, enabling on-demand access to adherence data. The next-generation Reader is a wrist-borne device.
  Other Names: Digital pill system
Drug: Truvada for pre-exposure prophylaxis (PrEP) — Participants will ingest one Truvada digital pill as PrEP per day, for 30 days total.
  Arms: PrEP Participants
Drug: Biktarvy for antiretroviral therapy (ART) — Participants will ingest one Biktarvy digital pill as ART per day, for 30 days total.
  Arms: ART Participants

SUMMARY:
This study will investigate the use of a next-generation Reader as part of a digital pill system (DPS; ID-Cap System) to measure adherence to both antiretroviral therapy (ART) and pre-exposure prophylaxis (PrEP) in people living with HIV (PLWH) and HIV-negative individuals, respectively. During the first (non-human subjects) component of this study, we developed a wrist-borne Reader according to design specifications and preferences shared by DPS users from our previous studies. Early bench testing by etectRx (manufacturer of the ID-Cap System) demonstrated that the wrist-borne version of the Reader acquires signal from the digital pill. This study will therefore evaluate the usability of and user response to a wrist-borne Reader component of the DPS among PLWH on ART and HIV-negative individuals on PrEP.

DETAILED DESCRIPTION:
This is a single-arm, observational trial (N=30), which will enroll N=15 people living with HIV (PLWH) using Biktarvy as antiretroviral therapy (ART) and N=15 HIV-negative individuals using Truvada as pre-exposure prophylaxis (PrEP). Potential participants will be approached and pre-screened. Those who meet pre-screening criteria will attend a Screening Visit (Visit 1), where the informed consent process will be conducted and eligibility will be confirmed. Eligible participants will attend a total of 3 study visits: the Screening Visit (Visit 1), Enrollment Visit (Visit 2), and Month 1 Visit (Visit 3). Participants will take one digital pill per day (Biktarvy as ART or Truvada as PrEP) for 30 days total, while using the next-generation Reader with a digital pill system, the ID-Cap System. Timeline followback discussions will be conducted at the Month 1 Visit to understand the context of any nonadherence detected by the digital pill system. Qualitative user experience exit interviews, quantitative assessments, dried blood spots (DBS), and pill counts of unused medication will also be conducted at the Month 1 Visit.

ELIGIBILITY:
Inclusion Criteria:

1. PrEP Participants:

   * Age 18 or older
   * HIV negative
   * Prescribed and currently taking Truvada for PrEP for at least 30 days
   * Qualifying labs for PrEP (Cr clearance in past 6 months, HBV vaccination, liver function tests)
   * Owns a smartphone with Android or iOS
2. ART Participants:

   * Age 18 or older
   * Diagnosed with HIV
   * Prescribed and taking Biktarvy for at least 6 months
   * Undetectable viral load during prior 6 months
   * Owns a smartphone with Android or iOS

Exclusion Criteria:

1. PrEP Participants:

   * Does not speak English
   * History of Crohn's disease or ulcerative colitis
   * History of gastric bypass or bowel stricture
   * History of GI malignancy or radiation to abdomen
   * Allergy to gelatin, silver, or zinc
   * Implanted cardiac device, nerve stimulator, or drug infusion pump
   * Not willing to operate DPS
2. ART Participants:

   * Does not speak English
   * History of Crohn's disease or ulcerative colitis
   * History of gastric bypass or bowel stricture
   * History of GI malignancy or radiation to abdomen
   * Allergy to gelatin, silver, or zinc
   * Implanted cardiac device, nerve stimulator, or drug infusion pump
   * Not willing to operate DPS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of Next-Generation ID-Cap System to Measure PrEP/ART Adherence | Month 1 study visit
  Participants' engagement with the digital pill system (DPS) -- the next-generation ID-Cap System -- will be measured over the 30-day study period. The percentages for the total expected ingestions recorded by the DPS each month will be compared to adherence detected by the DPS.
Correlation of PrEP/ART Adherence with DBS Concentrations and Pill Counts | Month 1 study visit
  Correlation of PrEP/ART adherence patterns, as detected by the next-generation ID-Cap System, with tenofovir diphosphate concentrations in dried blood spots (DBS) and pill counts of unused digital pills following the 30-day study period.
Acceptability of Next-Generation ID-Cap System, via System Usability Scale | Month 1 study visit
  Acceptability will be measured via the System Usability Scale (SUS). The SUS is a 10-item measure of perceived usability of a technological system, scored on a 5-point Likert scale (1: strongly disagree, 5: strongly agree), with higher scores indicating greater perceived usability. A mean score of >68 will be used to indicate that the technology is acceptable.
Acceptability of Next-Generation ID-Cap System, via Qualitative Interviews | Month 1 study visit
  Acceptability will be evaluated via qualitative interviews exploring participants' lived experiences operating the next-generation ID-Cap system and suggestions for improving the design of the technology.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chai, MD, MMS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Fenway Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No